CLINICAL TRIAL: NCT05847647
Title: Evaluation of the Effect of Leukocyte and Platelet-rich Fibrin on Clinical and Radiographic Healing After Periradicular Surgery: Randomized Controlled Clinical Trial.
Brief Title: Evaluation of the Effect of Leukocyte and Platelet-rich Fibrin on Healing After Periradicular Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seyda Ersahan, DDS, PhD (Other)
Responsible Party: Sponsor-Investigator, Seyda Ersahan, DDS, PhD, director, Istanbul Medipol University Hospital
Organization: Istanbul Medipol University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: periradicular surgery
Record Dates: First submitted 2023-02-01; First posted 2023-05-06 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Apical Periodontitis; Periapical Lesion
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1. group: Retrograde Filling Group / RG Group (Experimental): Surgical curettage of the periapical lesion and root tip resection will be performed, MTA will be applied retrogradely and no material will be applied to the bone defect
  Interventions: Other: Retrograde Filling Group
- 2. Group: Retrograde Filling+L-PRF Group / RG+L-PRF Group (Experimental): Surgical curettage of the periapical lesion and root tip resection will be performed, MTA will be applied retrogradely and L-PRF will be applied to the bone defect.
  Interventions: Other: Retrograde Filling+L-PRF Group
- 3. Group: Orthograde Filling Group / OG Group (Experimental): Surgical curettage of the periapical lesion will be performed, MTA will be applied orthogradely without root tip resection and no material will be applied to the bone defect.
  Interventions: Other: (Orthograde Filling Group / OG Group).
- 4. Group: Orthograde Filling+L-PRF Group / OG+L-PRF Group (Experimental): Surgical curettage of the periapical lesion will be performed, MTA will be applied orthogradely without root tip resection and L-PRF will be applied to the bone defect.
  Interventions: Other: (Orthograde Filling+L-PRF Group

INTERVENTIONS:
Other: Retrograde Filling Group — Surgical curettage of the periapical lesion and root tip resection will be performed, MTA will be applied retrogradely and no material will be applied to the bone defect.
  Arms: 1. group: Retrograde Filling Group / RG Group
Other: Retrograde Filling+L-PRF Group — 2. Group: Surgical curettage of the periapical lesion and root tip resection will be performed, MTA will be applied retrogradely and L-PRF will be applied to the bone defect (
  Arms: 2. Group: Retrograde Filling+L-PRF Group / RG+L-PRF Group
Other: (Orthograde Filling Group / OG Group). — 3. Group: Surgical curettage of the periapical lesion will be performed, MTA will be applied orthogradely without root tip resection and no material will be applied to the bone defect
  Arms: 3. Group: Orthograde Filling Group / OG Group
Other: (Orthograde Filling+L-PRF Group — 4. Group: Surgical curettage of the periapical lesion will be performed, MTA will be applied orthogradely without root tip resection and L-PRF will be applied to the bone defect
  Arms: 4. Group: Orthograde Filling+L-PRF Group / OG+L-PRF Group

SUMMARY:
The aim of this study is to evaluate the effect of two different periapical surgery methods ("curettage+apical resection" and "curettage") on the bone regeneration and clinical healing without applying any material or with applying leukocyte and platelet rich fibrin (L-PRF) to the periradicular intraosseous defect in the treatment of the teeth with large periapical lesions by following the patients for 12 months.

DETAILED DESCRIPTION:
Materials and Methods:

Apical periodontitis is a local response of the bone around the root tip of the tooth to necrosis of the pulp tissue. In the treatment of apical periodontitis, it is primarily aimed to remove the pathogenic microorganisms responsible for the infection with root canal treatment. The success of root canal treatment depends on the complete repair and regeneration of periapical tissues, and most of the periapical lesions heal satisfactorily after root canal treatment, but there are cases where infection and persistent symptoms persist despite root canal treatment. In these cases, periapical surgery with endodontic retreatment is required to eliminate pathological tissues, eliminate the source of irritation and support the healing process. For this purpose, 2 different periapical surgical methods are performed. In the first method, which is a more radical technique, the tip of the root of the related tooth responsible for apical periodontitis is resected (apicectomy) after curettage of the bone defect area. In the second method, in which the tooth tissue is preserved with a more conservative approach, only the defect area is curetted without root tip resection. Different results regarding the clinical success of these two methods have been reported in the literature.

In many studies, apicectomy is accepted as principal part of periapical surgical procedures and a prerequisite for the success of treatment but, roots that have already weakened and thinned due to periodontitis become more prone to fracture. In addition, especially in cases where the ratio between crown and root length is impaired, the stability of the restoration is adversely affected and the stability of the tooth in the socket may become questionable in the long term. In the literature, there are only a few case reports and a clinical study evaluating the clinical success of periapical surgery performed with periapical curettage without apicectomy following endodontic retreatment.

In recent years, many studies have been carried out to increase the success of apical surgery by accelerating and increasing the formation of new bone in the defect area with regenerative applications. Leukocyte and platelet-rich fibrin (L-PRF) is a second-generation platelet concentrate that forms an organized fibrin network in which platelets and leukocytes are trapped. In the few studies in the literature regarding the use of L-PRF alone without combining with a graft, in periapical surgery, apical surgery has been performed with root tip resection. In the literature, there is only one case series evaluating the effect of L-PRF application on periapical intraosseous defect after apical curettage without apicectomy on clinical and radiological healing.

In the treatment of apical periodontitis cases whith persistant symptoms and infection despite root canal treatment; more successful long-term results are aimed to be achieved by curettage of the periapical lesion and placement of L-PRF in the intraosseous defect after endodontic retreatment providing acceleration of apical bone regeneration, reducing clinical symptoms, and preserving the tooth root with a more conservative approach.

60 volunteer patients over the age of 18 who applied to Istanbul Medipol University Faculty of Dentistry, Department of Endodontics and were diagnosed with refractory chronic apical periodontitis due to a periapical lesion of endodontic origin that did not respond to root canal treatment, will be included in the study, regardless of gender. Periapical surgery will be applied in all patients following the endodontic retreatment.

Patients will be randomly divided into 4 groups of 15 patients in each group:

1. Group: Surgical curettage of the periapical lesion and root tip resection will be performed, MTA will be applied retrogradely and no material will be applied to the bone defect (Retrograde Filling Group / RG Group).
2. Group: Surgical curettage of the periapical lesion and root tip resection will be performed, MTA will be applied retrogradely and L-PRF will be applied to the bone defect (Retrograde Filling+L-PRF Group / RG+L-PRF Group).
3. Group: Surgical curettage of the periapical lesion will be performed, MTA will be applied orthogradely without root tip resection and no material will be applied to the bone defect (Orthograde Filling Group / OG Group).
4. Group: Surgical curettage of the periapical lesion will be performed, MTA will be applied orthogradely without root tip resection and L-PRF will be applied to the bone defect (Orthograde Filling+L-PRF Group / OG+L-PRF Group).

All surgical operations will be performed by the same surgeon, and all endodontic treatments will be performed by the same endodontist. Patients will be called for control for clinical and radiographic evaluation at 1. week and 1., 3., 6., 9., and 12. months. The PAI (Periapical index) score and the dimensions of the periapical radiolucency will be evaluated on the periapical radiographs taken at the control sessions. In addition, pain, swelling, tooth mobility, sensitivity to percussion, sensitivity of palpation and presence of fistula will be evaluated. Patients will be given forms including a 10-unit Numeric Rating Scale (NRS), and they will be asked to mark the pain they feel every day for 1 week postoperatively and to record the number of painkillers they use.

ELIGIBILITY:
60 volunteer patients over the age of 18 who applied to Istanbul Medipol University Faculty of Dentistry, Department of Endodontics and were diagnosed with refractory chronic apical periodontitis due to a periapical lesion of endodontic origin that did not respond to root canal treatment, will be included in the study, regardless of gender. Periapical surgery will be applied in all patients following the endodontic retreatment.

Inclusion Criteria:

1. Being over 18 years old.
2. systemic status is ASA I.
3. No history of allergy to local anesthetics and drugs to be used. D. Absence of a systemic disease or drug use that may adversely affect wound healing and contraindicate oral surgical procedures (radiotherapy, chemotherapy, corticosteroid use, antiplatelet or anticoagulant drug use, connective tissue diseases, vascular diseases, blood dyscrasia, liver diseases, uncontrolled diabetes, etc.).

to. Not smoking more than 10 cigarettes per day. f. Having a single rooted tooth of endodontic origin, with a periradicular lesion larger than 5 mm and smaller than 12 mm in diameter detected on periapical radiograph (chronic apical periodontitis), re-canal treatment planned and thought to be unsuccessful with re-canal treatment alone.

Exclusion Criteria:

1. Having ASA II-III-IV.
2. Having a history of allergy to local anesthetics and drugs to be used.
3. Presence of a systemic disease or drug use that may adversely affect postoperative wound healing and periodontal health.

D. Being pregnant or lactating. to. Not using antiplatelet or anticoagulant drugs and having blood dyscrasias f. Smoking more than 10 cigarettes per day. g. Vertical root fracture, perforation in the furcation region, endo-perio lesion and more than 5 mm periodontal bone loss in the involved tooth.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2024-09-02 (Estimated)

PRIMARY OUTCOMES:
Apical lesion healing | an average of 1 year
  Periapical index score and the dimensions of the periapical radiolucency will be evaluated on the periapical radiographs taken at the control sessions. In addition, pain, swelling, tooth mobility, sensitivity to percussion, sensitivity of palpation and presence of fistula will be evaluated.
  The PAI is a basic radiographic method of interpretation consisting of a scale from 1 to 5. It was first described by Ørstavik et al in 1986 (14). For each subject, the periapical tissue was assessed radiographically using the PAI as follows:
  1. PAI 1: normal periapical structure
  2. PAI 2: small changes in the bone structure not pathognomonic of apical periodontitis
  3. PAI 3: changes in the bone structure with mineral loss characteristic of apical periodontitis
  4. PAI 4: well-defined apical radiolucency characteristic of apical periodontitis
  5. PAI 5: severe periodontitis with exacerbating features and bone expansion

CONTACTS AND LOCATIONS:
Overall Officials: SEYDA ERSAHAN, Assoc.Prof., Study Director — Medipol University
Locations (1):
- Istanbul Medipol University, Faculty of Dentistry, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Gulsever S, Ersahan S, Hepsenoglu YE, Tekin A. Apicoectomy versus apical curettage in combination with or without L-PRF application: a randomized clinical trial. Sci Rep. 2025 Mar 8;15(1):8121. doi: 10.1038/s41598-025-92787-y. PMID 40057596